CLINICAL TRIAL: NCT02490137
Title: Brain Changes With Game Training in Aging
Acronym: BrainGame
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-1036
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Aging; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Game Players (Experimental): Participants that will play video game
  Interventions: Behavioral: Race Car Video Game
- Control (No Intervention): No video game experience

INTERVENTIONS:
Behavioral: Race Car Video Game — Repeatedly playing a race car video game
  Arms: Game Players

SUMMARY:
The purpose is to use MRI to investigate brain changes associated with playing a race car video game for 90 minutes in aging adults both with and without early signs of dementia.

DETAILED DESCRIPTION:
Neuroplasticity is an important process associated with memory and learning, and may be impaired in early Alzheimer's disease (AD). Video games are one potential strategy for investigating adaptive cognitive learning. Recent neuroimaging studies in healthy young adults have been able to detect brain changes associated with learning and memory from a racing video game over relatively short training periods of a couple hours. This strategy offers significant promise for characterizing the potential for neuroplasticity in patients at risk for AD including amnestic mild cognitive impairment (aMCI).

This project will apply video game training with magnetic resonance imaging (MRI) brain scanning to investigate adaptive learning, working memory and neuroplasticity as a function of aging and in patients with aMCI. A total of forty participants will be studied. Twenty subjects will undergo the video game training. Twenty subjects will be passive controls.

Specific Aims:

To characterize the microstructural brain changes after video game training in aging subjects and determine how patients with amnestic MCI (aMCI) and early AD are affected. For this study, adult participants ages 50 and older including patients with aMCI and early AD will undergo two neuroimaging sessions spaced roughly two hours apart that are bracketed around roughly 90 minutes of car racing game play. We will use diffusion-weighted imaging to detect longitudinal changes in microstructure of the hippocampus and parahippocampus. A primary objective of this study is to demonstrate that these training and imaging methods are translatable to patients with MCI. We will investigate the following two important hypotheses.

Hypothesis 1: Following car racing video game play, participants, on average, will demonstrate significant microstructural changes in hippocampal and parahippocampal brain regions measured with MRI.

Hypothesis 2: The microstructural changes in the hippocampus and parahippocampus measured with MRI will be significantly correlated with (a) cognitive memory performance as assessed by recent memory assessments, and (b) improvements in video game performance in all participants.

The primary outcome measures for both Hypotheses are the changes in the MRI measurements following car racing video game play.

A long-term objective of this project is to determine whether imaging short term neuroplasticity is predictive for individual patients of either future conversion to AD or the effectiveness of cognitive training therapies. More generally, neuroimaging markers of learning-induced brain plasticity would provide extremely useful tools for investigations of aging, dementias, and neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

1. 50-80 years of age
2. Part of existing aging research sample cohorts at University of Wisconsin - Madison
3. Successful research MRI study within prior two years
4. May include participants with

   1. No diagnosed cognitive impairment
   2. amnestic MCI
   3. mild AD (single or multi-domain) with predominant amnesia

Exclusion Criteria:

1. Contraindications to MRI (see Risks of MRI below)
2. Significant experience with playing race car video games in previous 2 years.
3. Severe AD
4. Lack of capacity as determined by the Capacity Assessment of Understanding questionnaire
5. Women who may be pregnant

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
MRI: Mean Diffusivity | 1.5-2 hours
  MRI based Mean Diffusivity changes in brain following playing video game for 90 minutes

SECONDARY OUTCOMES:
MRI: Structural Morphometry | 1.5-2 hours
  Local brain volumetric or shape changes

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Alexander, Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States